CLINICAL TRIAL: NCT00252655
Title: Use of Sirolimus Vs. Tacrolimus As The Primary Agent In Immunosuppressive Regimen For African-American Renal Allograft Recipients With Immediate Graft Function: A Pilot Study
Brief Title: Use of Sirolimus vs. Tacrolimus For African-American Renal Transplant Recipients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wayne State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 122102M1F
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Sirolimus; Tacrolimus

INTERVENTIONS:
Drug: Rapamune and Prograf

SUMMARY:
The purpose of this study is to evaluate the efficacy of Sirolimus (Rapamune) in improving the function of the transplant kidney, without any increase in the risk of acute rejection or adverse side effects, compared with Tacrolimus (Prograf).

We hypothesize that Sirolimus, as one component of a long-term steroid-free immunosuppressive regimen, will be effective in maintaining a low incidence of acute rejection and a short- and long-term graft survival comparable to Tacrolimus with better graft function in the high-risk African-American renal transplant population with immediate graft function.

DETAILED DESCRIPTION:
It has been repeatedly demonstrated that African-American renal allograft recipients have worse graft outcomes when compared with Caucasians. This has been attributed to various immunologic and non-immunologic factors, including a greater rate of acute rejection, resistance to standard doses of calcineurin inhibitors (CNIs) and corticosteroids, different pharmacokinetic and pharmacodynamic profiles, and noncompliance. It has therefore been suggested that quadruple immunosuppression, including antilymphocyte antibodies for induction, should be used in this high-risk population to improve graft survival. CNIs are currently the mainstay of immunosuppressive regimens. Tacrolimus has been shown to be significantly more effective than Cyclosporine A in preventing acute rejection. As a result, Tacrolimus has become the CNI of choice in preventing acute rejection, and has produced similar graft survival rates at one year, with higher creatinine clearances. However, there is no report examining the efficacy of Sirolimus in improving renal function and its side effect profile when compared with Tacrolimus in renal allograft recipients, particularly in African-Americans with immediate graft function in a steroid-free environment.

ELIGIBILITY:
Inclusion Criteria:

* African-American living- or deceased-donor renal transplant at least 18 years of age with current and historical negative crossmatch who demonstrate urine output > 60 ml/hr and fall in serum creatinine > 20%/day during the first 48 hours posttransplant, without need for dialysis.

Exclusion Criteria:

* Unwillingness to participate in the study
* Current PRA > 20%
* Noncompliance with the protocol and follow-up visits
* Those who need to be on maintenance steroids due to underlying disease
* Known hypersensitivity to study drugs
* Pregnancy
* Pre-transplant leukopenia, thrombocytopenia, hypercholesterolemia, or hypertriglyceridemia despite optimal medical therapy
* HIV positive recipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-01; Study Completion 2009-06

PRIMARY OUTCOMES:
Renal function at 1, 3, 6, and 12 months post transplant.

SECONDARY OUTCOMES:
Incidence of acute rejection.

CONTACTS AND LOCATIONS:
Overall Officials: Scott A. Gruber, MD, PhD, Principal Investigator — Harper University Hospital
Locations (1):
- Detroit Medical Center, Harper University Hospital, Detroit, Michigan, United States